CLINICAL TRIAL: NCT06641960
Title: The Effectiveness of Probiotics on Oral Health During Adult Orthodontic Treatment With Fixed Appliances: A Two-arm Parallel-group Randomized Controlled Clinical Trial
Brief Title: Using Probiotics to Improve Oral Hygiene During Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UDDS-Ortho-6-2024
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Orthodontic Appliance Complication
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Experimental): In this group, the patients will undergo orthodontic treatment with metallic appliances and receive oral hygiene instruction with probiotic lozenges.
  Interventions: Drug: Probiotics
- The control group without Probiotics (Active Comparator): In this group, the patients will undergo orthodontic treatment with metallic appliances and receive oral hygiene instruction without probiotic lozenges.
  Interventions: Procedure: Traditional treatment

INTERVENTIONS:
Drug: Probiotics — In this group, the patients will undergo orthodontic treatment with metallic appliances and receive oral hygiene instruction with probiotic lozenges.
  Arms: Probiotics group
Procedure: Traditional treatment — In this group, the patients will undergo orthodontic treatment with metallic appliances and receive oral hygiene instruction without probiotic lozenges.
  Arms: The control group without Probiotics

SUMMARY:
Fifty patients needing non-extraction-based metallic orthodontic treatment will be divided randomly into the probiotic group and the control group. In each group, they will brush their teeth regularly while receiving orthodontic treatment. Only the probiotic group will take probiotic tablets for six months.

Clinical parameters will be assessed before and during orthodontic treatment and after 3 and 6 months during treatment.

DETAILED DESCRIPTION:
Each subject will be examined completely to ensure eligibility before enrolling in the study. The operator will then inform them about the study's aim and ask them to provide written informed consent. Patients will receive professional scaling, polishing, and oral hygiene instruction before the research starts.

Regarding the probiotic, (PRODENTIS) is commercially available in Sweden and the USA. Probiotics prepared by Bio-Gaia AB (Stockholm, Sweden). Each probiotic tablet contains two strains of probiotic lactic acid bacteria of human origin: L. reuteri DSM 17938 and L. reuteri ATCC (PTA 5289), each at a minimum of 1 × 108 CFU per lozenge. The tablets should be stored at a temperature below 25 ◦C. Dosage instructions will be prescribed per the manufacturer's recommendations at a preventive dosage of 1 lozenge/day (after dinner and teeth brushing).

Regarding the clinical parameters, the Plaque index (Pl), the gingival index (GI), the Papillary Bleeding Index (PBI), 1977, and probing depth (PD) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy male and female patients aged 18-25 years.
2. Patients eligible for full arch upper and lower fixed labial orthodontic appliance treatment and molar band.
3. Patients with malocclusion class I, II, or III without crowding on the anterior teeth.
4. Permanent occlusion and existence of all the upper and lower teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Previous orthodontic treatment history.
2. Patients with any systemic disorder that could influence periodontal conditions or response to treatment (such as hypertension, diabetes, or immunological disorders).
3. Patients were on systemic drugs, i.e., antibiotics, hypertensives, analgesics, hormonal drugs, sedatives, and anti-seizure medication, within three months before the baseline examination.
4. Patients who were allergic to ingredients of the probiotics lozenges.
5. Those undergoing periodontal treatment within three months before the baseline examination.
6. Smokers, pregnant or lactating women.
7. Regular use of antibacterial mouthwash.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
The change in the plaque index | Time Frame: T0: immediately before applying the fixed appliance; T1: at three months; T2: at six months
  Assessment will be achieved using a gingival probe, according to Silness and Loe (1964). The criteria for plaque index are as follows:
  0. No plaque
  1. A film of plaque adheres to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after the application of the disclosing solution or by using a probe on the tooth surface.
  2. Moderate accumulation of soft deposits within the gingival pocket, or the tooth and the gingival margin, which can be seen with the naked eye.
  3. An abundance of soft matter within the gingival pocket and/or the tooth and gingival margin.
The change in the gingival index | Time Frame: T0: immediately before applying the fixed appliance; T1: at three months; T2: at six months
  Assessment will be achieved using a gingival probe, according to Silness and Loe (1964). The criteria for the gingival index are as follows:
  0. Normal gingiva.
  1. Mild inflammation: a slight change in color, slight edema, no bleeding on probing.
  2. Moderate inflammation: moderate glazing, redness, edema, hypertrophy, bleeding on probing.
  3. Severe inflammation: marked redness and hypertrophic ulceration, tendency to spontaneous bleeding.
The change in papillary bleeding index | Time Frame: T0: immediately before applying the fixed appliance; T1: at three months; T2: at six months
  Assessment will be achieved using a gingival probe, according to Muhlemann (1977).
  0. No bleeding.
  1. A single discreet bleeding point appears.
  2. Several isolated bleeding points or a single fine line of blood appear.
  3. The interdental triangle fills with blood shortly after probing.
  4. Profuse bleeding occurs after probing; blood flows immediately into the marginal sulcus.
The change in the probing depth | Time Frame: T0: immediately before applying the fixed appliance; T1: at three months; T2: at six months
  Assessment will be achieved using a gingival probe, according to Bowers (1964). It will be measured clinically as the distance from the free gingival margin to the gingival sulcus. The reading of PD ≤3 mm was considered normal, while any reading >3 mm was considered a gingival pocket

CONTACTS AND LOCATIONS:
Overall Officials: Lana Hasan Albardwel, DDS, Principal Investigator — Department of Orthodontics, Faculty of Dentistry, University of Damascus, Damascus , Syria
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damsacus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cerroni S, Pasquantonio G, Condo R, Cerroni L. Orthodontic Fixed Appliance and Periodontal Status: An Updated Systematic Review. Open Dent J. 2018 Sep 28;12:614-622. doi: 10.2174/1745017901814010614. eCollection 2018. PMID 30369970
- [Background] Contaldo M, Lucchese A, Lajolo C, Rupe C, Di Stasio D, Romano A, Petruzzi M, Serpico R. The Oral Microbiota Changes in Orthodontic Patients and Effects on Oral Health: An Overview. J Clin Med. 2021 Feb 16;10(4):780. doi: 10.3390/jcm10040780. PMID 33669186
- [Background] Agossa K, Dubar M, Lemaire G, Blaizot A, Catteau C, Bocquet E, Nawrocki L, Boyer E, Meuric V, Siepmann F. Effect of Lactobacillus reuteri on Gingival Inflammation and Composition of the Oral Microbiota in Patients Undergoing Treatment with Fixed Orthodontic Appliances: Study Protocol of a Randomized Control Trial. Pathogens. 2022 Jan 18;11(2):112. doi: 10.3390/pathogens11020112. PMID 35215057
- [Background] Freitas AO, Marquezan M, Nojima Mda C, Alviano DS, Maia LC. The influence of orthodontic fixed appliances on the oral microbiota: a systematic review. Dental Press J Orthod. 2014 Mar-Apr;19(2):46-55. doi: 10.1590/2176-9451.19.2.046-055.oar. PMID 24945514
- [Background] Santonocito S, Polizzi A. Oral Microbiota Changes during Orthodontic Treatment. Front Biosci (Elite Ed). 2022 Jul 27;14(3):19. doi: 10.31083/j.fbe1403019. PMID 36137992